CLINICAL TRIAL: NCT04782960
Title: The Effect of Subconjunctival Bupivacaine Injection in Squint Surgery for Postoperative Analgesia
Brief Title: Subconjunctival Bupivacaine in Strabismus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, abeer shaban, Lecture of Anesthesiology, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Subconjunctival bupivacaine
Record Dates: First submitted 2021-02-16; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia, Local
Keywords: Subconjunctival bupivacaine.; Strabismus surgery.; Postoperative analgesia.
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 patients receive Subconjunctival bupivacaine of the end of the surgery (Active Comparator): 20 patients receive Subconjunctival bupivacaine in the end of operation and monitoring postoperative pain score
  Interventions: Drug: Iocal anaesthetic bupivacaine
- 20 patients receive Subconjunctival placebo in the end of operation (Placebo Comparator): 20 patients receive Subconjunctival placebo in the end of operation and monitoring postoperative pain score
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iocal anaesthetic bupivacaine — Local anaesthetic Subconjunctival bupivacaine
  Other Names: Group (p)
  Arms: 20 patients receive Subconjunctival bupivacaine of the end of the surgery
Drug: Placebo — 0.9 saline
  Other Names: Group (s)
  Arms: 20 patients receive Subconjunctival placebo in the end of operation

SUMMARY:
This study aimed to assess the effectiveness of the Subconjunctival bupivacaine on postoperative pain in Strabismus surgery under general anaesthesia.

DETAILED DESCRIPTION:
40 patients will schedule for elective Strabismus surgery under general anaesthesia and randomly allocated into two groups to receive Subconjunctival 0.5%Bupivacaine group(B) or Subconjunctival placebo 0.9% normal saline group at the end of the surgery and assess the postoperative pain at 0th,30th, 60th,2nd h, 4h,6h,12h,24h.and post operative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 14 _30 years old with body mass index 18_28kg/m.
* American Anaesthesiologist Association physical states I,II.
* singed informed consent to participate in the study and were scheduled for strabismus operations under general anaesthesia.

Exclusion Criteria:

* were patients with chronic pain.
* ocular hypertension.
* inability to communicate.
* history of hematological disease.
* allergy to local anesthetic drugs.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) pain score | 5 minutes after extubation
  Range, 0_10;0,no pain ;10,worst pain

SECONDARY OUTCOMES:
Nausea and vomiting | 24 hours postoperatively
  Operation related side effect

OTHER OUTCOMES:
Patient satisfaction | 24 hours postoperatively
  Will be evaluated according to satisfaction score (poor=0, fair=1, good=2, excellent=3)
Visual analog scale (VAS) pain score | 30 minutes after extubation
  Range, 0_10;0,no pain ;10,worst pain
Visual analog scale (VAS) pain score | 60 minutes after extubation
  Range, 0_10;0,no pain ;10,worst pain
Visual analog scale (VAS) pain score | 2 hours after extubation
  Range, 0_10;0,no pain ;10,worst pain
Visual analog scale (VAS) pain score | 4 hours after extubation
  Range, 0_10;0,no pain ;10,worst pain
Visual analog scale (VAS) pain score | 6 hours after extubation
  Range, 0_10;0,no pain ;10,worst pain
Visual analog scale (VAS) pain score | 12 hours after extubation
  Range, 0_10;0,no pain ;10,worst pain
Visual analog scale (VAS) pain score | 24 hours after extubation
  Range, 0_10;0,no pain ;10,worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad A Hamed, MD, Study Director — Fayoum University Hospital

IPD SHARING:
Plan to Share IPD: No